CLINICAL TRIAL: NCT06848569
Title: Prospective, Single-Arm, Multicenter, Phase II Study of Sintilimab in Combination With AVD for Pediatric and Adolescent Low/Moderate Risk Classical Hodgkin Lymphoma
Brief Title: Sintilimab Plus AVD in Pediatric Low/Moderate Risk Hodgkin Lymphoma: A Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Prof, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-502-01
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab+AVD (Experimental)
  Interventions: Drug: Sintilimab in combination with AVD chemotherapy

INTERVENTIONS:
Drug: Sintilimab in combination with AVD chemotherapy — Sintilimab in combination with AVD chemotherapy treating classical Hodgkin lymphoma

SUMMARY:
Study Purpose: To evaluate the efficacy and safety of sintilimab in combination with AVD chemotherapy for the treatment of pediatric and adolescent patients with low-to-intermediate risk classical Hodgkin lymphoma (cHL).

Study Design: This is a prospective, single-arm, multicenter, phase II clinical trial.

Study Population: Pediatric and adolescent patients aged 1 to 18 years, diagnosed with classical Hodgkin lymphoma, and classified as low-to-intermediate risk according to the Ann Arbor staging system.

Treatment Plan: Sintilimab in combination with AVD chemotherapy, administered every two weeks for a planned 4-6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 and 18 years, regardless of gender.
2. Low-risk group: Must be a newly diagnosed patient with pathologically confirmed classical Hodgkin lymphoma, Ann Arbor stage IA or IIA, without bulky disease (defined as a mediastinal mass diameter > 1/3 of the chest diameter on an upright chest X-ray or any lymph node with a maximum transverse diameter > 6cm outside the mediastinum). Intermediate-risk group: Must be a newly diagnosed patient with pathologically confirmed classical Hodgkin lymphoma, Ann Arbor stage IB, IAE, IIAE, IIIA with or without bulky disease, or IA or IIA with bulky disease, or IIB without bulky disease (B symptoms defined as: weight loss > 10%; recurrent unexplained fever with temperature > 38°C; night sweats).
3. Presence of measurable lesions.
4. For male participants with reproductive potential, they must agree to the following during the intervention period to be eligible: not donating sperm, practicing abstinence according to their preferred and usual lifestyle, and agreeing to maintain abstinence or use contraception as required by the protocol unless proven to be azoospermic.
5. Female participants who are not pregnant or breastfeeding, non-reproductive potential women, or those who agree to use approved contraception for at least 120 days after the last research intervention, and agree not to donate eggs (ova, oocytes) to others or freeze/store for their own reproduction during this period.
6. General condition: Lansky score ≥ 50 (age < 16 years), Karnofsky score ≥ 50 (age ≥ 16 years).
7. Laboratory tests during the screening period should meet the following conditions:Absolute neutrophil count (ANC) ≥ 1.5×10^9/L (ANC ≥ 1.0×10^9/L if bone marrow involvement),Platelet count (PLT) ≥ 75×10^9/L (PLT ≥ 50×10^9/L if bone marrow involvement),Bilirubin ≤ 1.5 times the upper limit of normal (ULN) Creatinine ≤ 1.5 times ULN (calculated according to the standard Cockcroft-Gault formula).ALT/AST ≤ 3 times ULN (can be relaxed to 5 times ULN if liver metastasis is present)
8. Able to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits during participation in the study.
9. Parents/legal guardians of pediatric or adolescent subjects have the ability to understand, consent, and sign the informed consent form (ICF) and applicable child assent form before any protocol-related procedures are initiated; subjects are able to express consent in the presence of parents/legal guardians (if applicable).

Exclusion Criteria:

1. History of solid organ transplantation at any time or allogeneic hematopoietic stem cell transplantation within the past 5 years.
2. Female participants with reproductive potential who test positive for pregnancy on a urine pregnancy test within 24 hours before the first dose.
3. Baseline left ventricular ejection fraction < 50% or left ventricular short-axis shortening fraction < 27%.
4. Previous treatment with anti-programmed death (PD-1), anti-programmed death ligand 1 (PD-L1), or anti-PD-L2 drugs, or drugs targeting another co-inhibitory T cell receptor.
5. Received any systemic anti-cancer treatment, including investigational drugs for the current diagnosis, before enrollment.
6. Received live or attenuated vaccines within 30 days before the first research intervention. Inactivated vaccines are allowed.
7. Received investigational drugs or used investigational devices within 4 weeks before the research intervention.
8. Diagnosed with lymphocyte-predominant Hodgkin lymphoma.
9. Diagnosed with immune deficiency or receiving chronic systemic corticosteroid therapy or any other form of immunosuppressive treatment within 7 days before the first administration of sintilimab.
10. Known progression of other malignancies or requiring active treatment within the past 3 years.
11. Presence of detectable central nervous system metastasis and/or carcinomatous meningitis on radiology at the time of diagnosis.
12. Severe hypersensitivity (≥ grade 3) to any research treatment, including excipients.
13. Active autoimmune disease requiring systemic treatment within the past 2 years.
14. History of (non-infectious) pneumonia/interstitial pneumonitis requiring corticosteroid treatment or currently suffering from pneumonia/interstitial lung disease with active infection requiring systemic treatment.
15. Known history of human immunodeficiency virus (HIV) infection.
16. Known history of hepatitis B or active hepatitis C virus infection.
17. Presence of any disease, treatment, or laboratory abnormality results that may confound study results, interfere with the subject's participation throughout the study, or, in the opinion of the treating investigator, is not in the subject's best interest to participate in the study.
18. Known mental illness or substance abuse disorder that would interfere with cooperation with the study requirements.
19. Patient has not fully recovered from major surgery or has persistent postoperative complications.
20. Other conditions that the investigator considers should be excluded.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-10-23 (Estimated); Study Completion 2031-10-23 (Estimated)

PRIMARY OUTCOMES:
4-year event-free survival | 4 years
  The 4-year event-free survival (EFS) rate of pediatric and adolescent patients with low-to-intermediate risk classical Hodgkin lymphoma (cHL) treated with sintilimab in combination with the AVD regimen. EFS is defined as the time from study entry to the occurrence of disease progression, relapse, second primary malignancy, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China